CLINICAL TRIAL: NCT06454578
Title: An Open-Label, Single Arm Study to Evaluate the Efficacy and Safety of Adebrelimab Plus Apatinib as Adjuvant Therapy in Participants With Hepatocellular Carcinoma at High Risk of Recurrence After Surgical Resection
Brief Title: Adjuvant Adebrelimab Plus Apatinib for Participants With HCC at High-risk of Recurrence After Curative Resection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202401-002-1
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab + Apatinib (Experimental)
  Interventions: Drug: Adebrelimab + Apatinib

INTERVENTIONS:
Drug: Adebrelimab + Apatinib — the first 6 months or 8 cycles: Adebrelimab 1200 mg, every 3 weeks； Apatinib 250 mg/day
  Maintenance phase： Adebrelimab 1200 mg, every 3 weeks, Maximum maintenance up to 2 years

SUMMARY:
This is a single-center, single-arm, open-label clinical study to evaluate the efficacy and safety of Adebrelimab plus Apatinib as adjuvant therapy in hepatocellular carcinoma (HCC) participants who are at high risk of recurrence after curative resection.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a malignant tumor with high morbidity and mortality. Surgical resection is the most important radical treatment. However, the recurrence rate is high especially in the participants with high risk of recurrence after curative resection.

Adebelimumab is a humanized anti-PD-L1 monoclonal antibody independently developed by Hengrui Pharmaceutical. It can specifically bind to PD-L1 molecules to block the PD-1/PD-L1 pathway that leads to tumor immune tolerance, reactivate the anti-tumor activity of the immune system, and achieve the goal of treating tumors. As of October 8, 2021, adebelimumab has conducted several clinical studies in various malignant tumor fields and has shown good anti-tumor efficacy and controllable safety.

Therefore, the investigators plan to conduct a prospective clinical study targeting HCC participants at high risk of postoperative recurrence, to demonstrate the efficacy and safety of postoperative adjuvant therapy with adebelimumab combined with apatinib. This study has the potential to provide efficient new treatment options for participants, which is of great significance for improving the survival rate and quality of life of liver cancer participants in general.

A mid-term analysis will be conducted on the recurrence free survival rate and survival rate, at 6 months after the enrollment of 30 participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following conditions in order to be enrolled in this study:

1. Voluntarily participate in this study and sign an informed consent form.
2. Participants diagnosed with HCC through pathological histology/cytology or clinically diagnosed with HCC according to the Diagnosis and Treatment Guidelines for Primary Liver Cancer (2024 Edition).
3. Within 4-12 weeks prior to enrollment, radical resection surgery was performed.
4. Complete recovery from surgical resection within 4 weeks prior to enrollment.
5. High risk factors for postoperative recurrence of hepatocellular carcinoma include multiple tumors, tumor length>5 cm, poor tumor differentiation (Edmondson III-IV grade), margin ≤ 1 cm, invasion of Microvasculature or large vessels, lymph node metastasis, sustained abnormalities in AFP or abnormal prothrombin , etc.
6. Child Pugh liver function rating within 7 days prior to randomization: A or B (≤ 7 points).
7. ECOG PS score within 7 days before randomization: 0-1 points.
8. Have not received systematic anti-tumor treatment for hepatocellular carcinoma in the past.
9. Expected survival time ≥ 12 weeks.
10. The main organ functions meet the following requirements (within 7 days before randomization):

(1) Blood routine examination: (excluding hemoglobin, no blood transfusion within 14 days prior to screening, no use of granulocyte colony-stimulating factor [G-CSF], no medication correction):

• Neutrophil absolute count ≥ 1.5 × 109/L; Platelets ≥ 75 × 10^9/L; • Hemoglobin ≥ 90 g/L.(Leukocyte and thrombocytopenia caused by splenic hyperfunction can be included in the group after partial embolization of the splenic artery or medication correction) (2) Blood biochemistry test (no albumin transfusion within 14 days before screening): Serum albumin ≥ 28g/L; Total serum bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN; Blood creatinine ≤ 1.5 x ULN or Cr clearance rate>50ml/min (3) International standardized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeding the range of normal control ≤ 6 (4) Urinary protein<2+(If urinary protein ≥ 2+, 24-hour urine protein quantification is required, and 24-hour urine protein quantification<1.0g can be included in the group).

11. If suffering from hepatitis B virus (HBV) infection, it is necessary to be willing to receive antiviral treatment throughout the study period (according to the diagnostic and treatment guidelines, such as entecavir) and regularly monitor it; Hepatitis C virus (HCV) ribonucleic acid (RNA) positive subjects must receive antiviral treatment according to the diagnosis and treatment guidelines, and their liver function must be within CTCAE1 level elevation.

12.Women with fertility: must agree to contraception from the signing of the informed consent form until 90 days after the last use of the study drug (whichever is longer). And the blood HCG test must be negative within 7 days before starting the study treatment; And it must be non lactation period

Exclusion Criteria:

If a subject meets any of the following conditions, they will not be allowed to enter this study:

1. Known hepatobiliary carcinoma, sarcoma like hepatocellular carcinoma, combined hepatocellular-cholangiocarcinoma，and fibrous layer cell carcinoma; Within 5 years or simultaneously suffering from other active malignant tumors other than hepatocellular carcinoma (excluding cured skin basal cell carcinoma and cervical carcinoma in situ).
2. There are uncontrollable extrahepatic metastases, such as lung and brain metastases (EHS).
3. Previously received local treatment, including therapeutic TACE, transarterial embolization (TAE), hepatic artery infusion chemotherapy (HAIC), transarterial radiation embolization (TARE), etc.
4. Participants who are preparing to undergo or have previously received organ or allogeneic bone marrow transplantation.
5. Participants who are currently accompanied by interstitial pneumonia or interstitial lung disease, or have a history of interstitial pneumonia or interstitial lung disease that requires hormone therapy in the past, or other pulmonary fibrosis, organized pneumonia (such as bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or subjects with evidence of active pneumonia or severe lung function impairment seen on chest computed tomography (CT) images during screening, are allowed to have radiation induced pneumonia in the radiation field; Active tuberculosis.
6. Currently, there is active autoimmune disease or a history of autoimmune disease that may recur (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects that can be controlled only through hormone replacement therapy can be included]); Subjects with skin diseases that do not need systematic treatment, such as vitiligo, psoriasis, alopecia, controlled type I diabetes that receive insulin treatment, or childhood asthma that has completely alleviated without any intervention after adulthood can be included; Asthma subjects who require medical intervention with bronchodilators cannot be included.
7. Suffering from hypertension and unable to achieve good control through antihypertensive drug treatment (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg) (based on the average BP reading obtained from ≥ 2 measurements), it is allowed to achieve the above parameters through the use of antihypertensive therapy; Previously experienced hypertensive crisis or hypertensive encephalopathy.
8. Participants with moderate to severe ascites with clinical symptoms who require therapeutic puncture or drainage, or whose Child Pugh score is greater than 7 (excluding those who only show a small amount of ascites on imaging but do not have clinical symptoms); Uncontrolled or moderate to equal amounts of pleural effusion and pericardial effusion.
9. There are clinical symptoms or diseases of the heart that cannot be well controlled, such as: (1) According to the standards of the New York Heart Association (NYHA), level II or above cardiac insufficiency or cardiac ultrasound examination: LVEF (left ventricular ejection fraction)<50%; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year prior to the start of the research treatment; (4) Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention; (5) QTc>480ms (QTc interval is calculated using the Fridericia formula; if QTc is abnormal, it can be detected continuously three times every 2 minutes, and the average value is taken).
10. History of spontaneous rupture of liver tumors.
11. Individuals with a history of hepatic encephalopathy.
12. Congenital or acquired immune dysfunction in subjects (such as HIV infected individuals).
13. There have been incidents of thrombosis or embolism occurring within the first 6 months of treatment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
14. Participants with a history of gastrointestinal bleeding or a clear tendency towards gastrointestinal bleeding within 6 months prior to the start of the study treatment, such as those at risk of bleeding or severe esophageal and gastric varices, locally active gastrointestinal ulcer lesions, or continuous positive fecal occult blood, cannot be included in the study. (If fecal occult blood is positive during the baseline period, a follow-up examination is required. If the follow-up examination is still positive, gastroduodenoscopy (EGD) is required. If EGD indicates a risk of bleeding, esophageal and gastric varices/other gastrointestinal diseases cannot be included in the study.)
15. Within 6 months prior to the start of treatment, there have been abdominal fistulas, gastrointestinal perforation, or abdominal abscesses.
16. Severe, unhealed or cracked wounds, as well as active ulcers or untreated fractures.
17. Known genetic or acquired bleeding (such as coagulation dysfunction) or thrombotic tendencies, such as in hemophilia participants; Currently or recently (within 10 days prior to the start of research treatment), full dose oral or injection anticoagulants or thrombolytic drugs (prophylactic use of low-dose aspirin, low molecular weight heparin allowed) have been used for therapeutic purposes.
18. Major vascular diseases (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) occur within 6 months prior to the start of the study treatment.
19. Severe infection within 4 weeks prior to the start of the study treatment, including but not limited to hospitalization due to complications of infection, bacteremia, or severe pneumonia; Oral or intravenous administration of therapeutic antibiotics within 2 weeks prior to the start of the study treatment (subjects who receive prophylactic antibiotics, such as preventing urinary tract infections or exacerbation of chronic obstructive pulmonary disease, are eligible to participate in the study).
20. It is known that the active ingredients and excipients contained in the investigational drugs (Adebelimumab, Apatinib) in this study have hypersensitivity reactions, or have a history of severe allergies to any other monoclonal antibodies or anti angiogenic targeted drugs.
21. Use immunosuppressive agents or systemic hormone therapy within 14 days prior to the start of the study to achieve immunosuppressive effects (dose>10mg/day prednisone or other therapeutic hormones).
22. Received attenuated live vaccine treatment within 28 days prior to the start of the study treatment, or expected to receive such vaccines during the treatment period with Adebrelimab or within 60 days after the last dose of Adebrelimab.
23. Received other experimental drug treatments within 28 days or 5 half-lives (whichever is longer) prior to the start of the study treatment.
24. According to the judgment of the researchers, the subjects may have other factors that may affect the research results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious illnesses (including mental illness) that require concurrent treatment, serious laboratory test abnormalities, and family or social factors that may affect the safety of the subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
RFS Rate at 12 and 24 Months | up to 24 months
  Recurrence-free survival rate at 12 and 24 Months

SECONDARY OUTCOMES:
overall survival | 3 years
  Defined as the time from enrollment to death from any cause
Time to Recurrence | up to 3 years
  The time interval between liver resection and diagnosis of HCC recurrence
recurrence-free survival | up to 3 years
  Ratio of participants from first treatment to disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Tao Li, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China